CLINICAL TRIAL: NCT02114268
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Dose-escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MEDI8897 in Healthy Adults
Brief Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MEDI8897 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D5290C00001
Record Dates: First submitted 2014-04-03; First posted 2014-04-15 (Estimated); Results first posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus, RSV
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- MEDI8897 300 milligram (mg) Intravenous (IV) (Experimental): Participants received a single fixed dose of 300 mg MEDI8897 intravenous infusion on Day 1.
  Interventions: Drug: MEDI8897 Intravenous
- MEDI8897 1000 mg IV (Experimental): Participants received a single fixed dose of 1000 mg MEDI8897 intravenous infusion on Day 1.
  Interventions: Drug: MEDI8897 Intravenous
- MEDI8897 3000 mg IV (Experimental): Participants received a single fixed dose of 3000 mg MEDI8897 intravenous infusion on Day 1.
  Interventions: Drug: MEDI8897 Intravenous
- MEDI8897 100 mg Intramuscular (IM) (Experimental): Participants received a single fixed dose of 100 mg MEDI8897 intramuscular injection on Day 1.
  Interventions: Drug: MEDI8897 Intramuscular
- MEDI8897 300 mg IM (Experimental): Participants received a single fixed dose of 300 mg MEDI8897 intramuscular injection on Day 1.
  Interventions: Drug: MEDI8897 Intramuscular
- Placebo (Placebo Comparator): Participants received placebo on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEDI8897 Intravenous — Participants received a single fixed dose of 300 mg MEDI8897 intravenous infusion on Day 1.
  Arms: MEDI8897 300 milligram (mg) Intravenous (IV)
Drug: Placebo — Participants received placebo on Day 1.
  Arms: Placebo
Drug: MEDI8897 Intravenous — Participants received a single fixed dose of 1000 mg MEDI8897 intravenous infusion on Day 1.
  Arms: MEDI8897 1000 mg IV
Drug: MEDI8897 Intravenous — Participants received a single fixed dose of 3000 mg MEDI8897 intravenous infusion on Day 1.
  Arms: MEDI8897 3000 mg IV
Drug: MEDI8897 Intramuscular — Participants received a single fixed dose of 100 mg MEDI8897 intramuscular injection on Day 1.
  Arms: MEDI8897 100 mg Intramuscular (IM)
Drug: MEDI8897 Intramuscular — Participants received a single fixed dose of 300 mg MEDI8897 intramuscular injection on Day 1.
  Arms: MEDI8897 300 mg IM

SUMMARY:
The purpose of this study was to evaluate the safety, tolerability and pharmacokinetics of an extended half-life anti-respiratory syncytial virus (RSV) monoclonal antibody compared to placebo when administered to healthy adult participants.

DETAILED DESCRIPTION:
This was a phase 1, randomized, double-blind, placebo-controlled, dose-escalation study to evaluate the safety, tolerability and pharmacokinetics of MEDI8897 compared to placebo when administered to healthy adult participants. There were 136 participants randomized to receive MEDI8897 or placebo at one site. Investigational product was delivered intravenously (IV) to 3 cohorts and intramuscularly (IM) to 2 cohorts. 4 different dose levels of investigational product were evaluated across the 5 cohorts. Participants were followed for approximately 1 year.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 18 through 49 years and in good health by history, physical exam, and labs
* Weight greater than or equal to (>=) 45 kilogram (kg) and less than or equal to (<=) 110 kg at Screening
* Written informed consent prior to performing any protocol related procedures, including Screening evaluations
* Ability to complete the Follow-up period of 360 days

Key Exclusion Criteria:

* Acute illness including fever >= 99.5 Fahrenheit (°F) on day of dosing
* Any drug therapy within 7 days prior to Day 1 (except contraceptives)
* Receipt of any investigational drug therapy within 120 days prior to investigational product dosing through 360 days after investigational product dosing
* Previous receipt of a monoclonal antibody (mAb)
* Pregnant or nursing mother
* Concurrent enrollment in another interventional study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 342 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Pamela Griffin, MD, Study Director — MedImmune LLC; Martin Kankam, MD, PhD, MPH, Principal Investigator — Study Site
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Griffin MP, Khan AA, Esser MT, Jensen K, Takas T, Kankam MK, Villafana T, Dubovsky F. Safety, Tolerability, and Pharmacokinetics of MEDI8897, the Respiratory Syncytial Virus Prefusion F-Targeting Monoclonal Antibody with an Extended Half-Life, in Healthy Adults. Antimicrob Agents Chemother. 2017 Feb 23;61(3):e01714-16. doi: 10.1128/AAC.01714-16. Print 2017 Mar. PMID 27956428

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 342 participants who were screened. A total of 136 participants met eligibility criteria and were randomized into the study.
Groups:
- MEDI8897 300 Milligram (mg) Intravenous (IV): Participants received single fixed dose of 300 mg MEDI8897 intravenous infusion on Day 1.
- MEDI8897 1000 Milligram (mg) Intravenous (IV): Participants received single fixed dose of 1000 mg MEDI8897 intravenous infusion on Day 1.
- MEDI8897 3000 Milligram (mg) Intravenous (IV): Participants received single fixed dose of 3000 mg MEDI8897 intravenous infusion on Day 1.
- MEDI8897 100 Milligram (mg) Intramuscular (IM): Participants received single fixed dose of 100 mg MEDI8897 intramuscular injection on Day 1.
- MEDI8897 300 Milligram (mg) Intramuscular (IM): Participants received single fixed dose of 300 mg MEDI8897 intramuscular injection on Day 1.
Period: Overall Study
Arm/Group | Placebo | MEDI8897 300 Milligram (mg) Intravenous (IV) | MEDI8897 1000 Milligram (mg) Intravenous (IV) | MEDI8897 3000 Milligram (mg) Intravenous (IV) | MEDI8897 100 Milligram (mg) Intramuscular (IM) | MEDI8897 300 Milligram (mg) Intramuscular (IM)
Started | 34 | 6 | 6 | 6 | 6 | 78
Completed | 28 | 5 | 5 | 6 | 6 | 75
Not Completed | 6 | 1 | 1 | 0 | 0 | 3
Not completed — Lost to Follow-up | 4 | 1 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawn by site due to noncompliance | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The As-treated Population included participants who receive any study investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI8897 300 Milligram (mg) Intravenous (IV) | MEDI8897 1000 Milligram (mg) Intravenous (IV) | MEDI8897 3000 Milligram (mg) Intravenous (IV) | MEDI8897 100 Milligram (mg) Intramuscular (IM) | MEDI8897 300 Milligram (mg) Intramuscular (IM) | Total
Number analyzed (Participants) | 34 | 6 | 6 | 6 | 6 | 78 | 136
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.2 (8.6) | 34.5 (8.6) | 34.3 (5.6) | 33.5 (6.7) | 30.7 (7.8) | 30.3 (7.9) | 30.5 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 4 | 2 | 3 | 6 | 39 | 73
  Male | 15 | 2 | 4 | 3 | 0 | 39 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is defined as events present at baseline that worsened in intensity after administration of investigational products or events absent at baseline that emerged after administration of study drug, for the period extending to 391 (Day 361 ± 30 days) days after the last dose of study drug.
Time Frame: From start of study drug administration up to Day 391 (Day 361 +/- 30 days)
Population: The As-treated population included participants who receive any study investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | MEDI8897 300 Milligram (mg) Intravenous (IV) | MEDI8897 1000 Milligram (mg) Intravenous (IV) | MEDI8897 3000 Milligram (mg) Intravenous (IV) | MEDI8897 100 Milligram (mg) Intramuscular (IM) | MEDI8897 300 Milligram (mg) Intramuscular (IM)
Number analyzed (Participants) | 34 | 6 | 6 | 6 | 6 | 78
participants
  TEAEs | 21 | 3 | 3 | 5 | 4 | 48
  TESAEs | 0 | 0 | 0 | 0 | 0 | 2

2. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of MEDI8897
Description: The Tmax is defined as actual sampling time to reach maximum observed MEDI8897 concentration. The reported Standard Deviation values are actually Relative Standard Deviation (RSD) values (that is, Coefficient of Variation).
Time Frame: Predose, End of Dosing (IV Arms), 8 Hour Postdose, Day 2, 4, 6, 8, 15, 22, 31, 61, 91, 121, 151, 181, 271 and 361
Population: Pharmacokinetic parameter analysis population included all randomized population treated with MEDI8897. Number of participants analyzed signifies those participants who were evaluable for the measure.
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | MEDI8897 300 Milligram (mg) Intravenous (IV) | MEDI8897 1000 Milligram (mg) Intravenous (IV) | MEDI8897 3000 Milligram (mg) Intravenous (IV) | MEDI8897 100 Milligram (mg) Intramuscular (IM) | MEDI8897 300 Milligram (mg) Intramuscular (IM)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 78
Day | 0.078 (172) | 0.059 (0) | 0.209 (62.7) | 5.46 (71.4) | 9.42 (78.4)

3. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for MEDI8897
Description: The Cmax is the maximum observed serum concentration of MEDI8897. The reported Standard Deviation values are actually Relative Standard Deviation (RSD) values (that is, Coefficient of Variation).
Time Frame: Predose, End of Dosing (IV Arms), 8 Hour Postdose, Day 2, 4, 6, 8, 15, 22, 31, 61, 91, 121, 151, 181, 271 and 361
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/ml)
Arm/Group | MEDI8897 300 Milligram (mg) Intravenous (IV) | MEDI8897 1000 Milligram (mg) Intravenous (IV) | MEDI8897 3000 Milligram (mg) Intravenous (IV) | MEDI8897 100 Milligram (mg) Intramuscular (IM) | MEDI8897 300 Milligram (mg) Intramuscular (IM)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 78
microgram per milliliter (mcg/ml) | 96.98 (21.9) | 333.80 (22.4) | 1163.32 (23.8) | 20.40 (29.4) | 47.48 (26.2)

4. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) for MEDI8897
Description: The AUC (0-infinity) is the area under the serum concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the serum concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant. The reported Standard Deviation values are actually Relative Standard Deviation (RSD) values (that is, Coefficient of Variation).
Time Frame: Predose, End of Dosing (IV Arms), 8 Hour Postdose, Day 2, 4, 6, 8, 15, 22, 31, 61, 91, 121, 151, 181, 271 and 361
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Day*microgram per milliliter
Arm/Group | MEDI8897 300 Milligram (mg) Intravenous (IV) | MEDI8897 1000 Milligram (mg) Intravenous (IV) | MEDI8897 3000 Milligram (mg) Intravenous (IV) | MEDI8897 100 Milligram (mg) Intramuscular (IM) | MEDI8897 300 Milligram (mg) Intramuscular (IM)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 75
Day*microgram per milliliter | 6714.75 (21.7) | 25320.68 (17) | 63580.33 (10.4) | 2249.11 (17.9) | 5193.73 (32.1)

5. Secondary Outcome: Terminal Phase Elimination Half Life (t1/2) for MEDI8897
Description: The terminal elimination half-life (t1/2) is the time measured for the serum concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z). Here 'n' signifies participants evaluable for specified categories, for each arm, respectively. The reported Standard Deviation values are actually Relative Standard Deviation (RSD) values (that is, Coefficient of Variation).
Time Frame: Predose, End of Dosing (IV Arms), 8 Hour Postdose, Day 2, 4, 6, 8, 15, 22, 31, 61, 91, 121, 151, 181, 271 and 361
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | MEDI8897 300 Milligram (mg) Intravenous (IV) | MEDI8897 1000 Milligram (mg) Intravenous (IV) | MEDI8897 3000 Milligram (mg) Intravenous (IV) | MEDI8897 100 Milligram (mg) Intramuscular (IM) | MEDI8897 300 Milligram (mg) Intramuscular (IM)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 75
Day | 116.52 (19.6) | 92.0 (12.6) | 89.81 (18.2) | 102.61 (11.3) | 85.29 (30.8)

6. Secondary Outcome: Systemic Clearance (CL) for MEDI8897
Description: Systemic Clearance (CL) is a quantitative measure of the rate at which a drug substance is removed from the body. The total systemic clearance after the dose was estimated by dividing the total administered dose by the Area Under the Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]). Apparent clearance (CL/F) for the IM dose groups. The reported Standard Deviation values are actually Relative Standard Deviation (RSD) values (that is, Coefficient of Variation).
Time Frame: Predose, End of Dosing (IV Arms), 8 Hour Postdose, Day 2, 4, 6, 8, 15, 22, 31, 61, 91, 121, 151, 181, 271 and 361
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml per day
Arm/Group | MEDI8897 300 Milligram (mg) Intravenous (IV) | MEDI8897 1000 Milligram (mg) Intravenous (IV) | MEDI8897 3000 Milligram (mg) Intravenous (IV) | MEDI8897 100 Milligram (mg) Intramuscular (IM) | MEDI8897 300 Milligram (mg) Intramuscular (IM)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 75
ml per day | 46.05 (17.3) | 40.33 (15.4) | 47.60 (10.6) | 45.46 (15.4) | 64.60 (37.7)

7. Secondary Outcome: Volume of Distribution (Vz) for MEDI8897
Description: The Vz is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a study drug. Apparent volume of distribution (Vz/F) for the IM dose groups. The reported Standard Deviation values are actually Relative Standard Deviation (RSD) values (that is, Coefficient of Variation).
Time Frame: Predose, End of Dosing (IV Arms), 8 Hour Postdose, Day 2, 4, 6, 8, 15, 22, 31, 61, 91, 121, 151, 181, 271 and 361
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliter (ml)
Arm/Group | MEDI8897 300 Milligram (mg) Intravenous (IV) | MEDI8897 1000 Milligram (mg) Intravenous (IV) | MEDI8897 3000 Milligram (mg) Intravenous (IV) | MEDI8897 100 Milligram (mg) Intramuscular (IM) | MEDI8897 300 Milligram (mg) Intramuscular (IM)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 75
milliliter (ml) | 7694.15 (24.8) | 5426.89 (26.7) | 6137.69 (18.5) | 6808.78 (24.5) | 7455.90 (34.0)

8. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA)
Description: Participants were tested for anti-drug antibody to MEDI8897 prior to enrollment, predose and postdose.
Time Frame: Predose and Day 15, 31, 91, 181, 271 and 361
Population: The As-treated Population included participants who receive any study investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | MEDI8897 300 Milligram (mg) Intravenous (IV) | MEDI8897 1000 Milligram (mg) Intravenous (IV) | MEDI8897 3000 Milligram (mg) Intravenous (IV) | MEDI8897 100 Milligram (mg) Intramuscular (IM) | MEDI8897 300 Milligram (mg) Intramuscular (IM)
Number analyzed (Participants) | 34 | 6 | 6 | 6 | 6 | 78
participants
  Predose | 3 | 0 | 0 | 0 | 0 | 5
  At Any Time Postdose | 5 | 0 | 1 | 0 | 0 | 13

ADVERSE EVENTS:
Time Frame: From Screening to Postdose Follow-up (up to 391 Days)
Arm/Group | Placebo | MEDI8897 300 Milligram (mg) Intravenous (IV) | MEDI8897 1000 Milligram (mg) Intravenous (IV) | MEDI8897 3000 Milligram (mg) Intravenous (IV) | MEDI8897 100 Milligram (mg) Intramuscular (IM) | MEDI8897 300 Milligram (mg) Intramuscular (IM)
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/6 | 0/6 | 0/6 | 0/6 | 2/78
Other Adverse Events (participants affected / at risk) | 21/34 | 3/6 | 3/6 | 5/6 | 4/6 | 48/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=34) | MEDI8897 300 Milligram (mg) Intravenous (IV) (N=6) | MEDI8897 1000 Milligram (mg) Intravenous (IV) (N=6) | MEDI8897 3000 Milligram (mg) Intravenous (IV) (N=6) | MEDI8897 100 Milligram (mg) Intramuscular (IM) (N=6) | MEDI8897 300 Milligram (mg) Intramuscular (IM) (N=78)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=34) | MEDI8897 300 Milligram (mg) Intravenous (IV) (N=6) | MEDI8897 1000 Milligram (mg) Intravenous (IV) (N=6) | MEDI8897 3000 Milligram (mg) Intravenous (IV) (N=6) | MEDI8897 100 Milligram (mg) Intramuscular (IM) (N=6) | MEDI8897 300 Milligram (mg) Intramuscular (IM) (N=78)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Salivary gland pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug intolerance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 16 (19)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 7 (8)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polycystic ovaries (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Physical examination parameters of participants were not evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.